CLINICAL TRIAL: NCT02133807
Title: A 72-week, Prospective, Parallel-group, Partially Blinded, Controlled Phase IIIb Study Evaluating the Impact of Specific Lp(a) Apheresis on Atherosclerotic Disease Burden in Coronary Heart Disease Patients With High Lipoprotein(a) Level.
Brief Title: Specific Lp(a) Apheresis for Regression of Coronary and Carotid Atherosclerosis
Acronym: LaRCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Russian Cardiology Research and Production Center (Other)
Collaborators: Clinical Diagnostic Center MEDSI (Unknown); Moscow State Government (Unknown)
Responsible Party: Principal Investigator, Professor Sergei Pokrovsky, PhD, DSc, Chair of the Laboratory of Atherosclerosis, Russian Cardiology Research and Production Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01200953720
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Atherosclerosis; Coronary Disease; Carotid Artery Diseases
Keywords: Lipoprotein(a);; Lp(a) immunoadsorption;; Apheresis;; Coronary atherosclerosis;; Carotid Atherosclerosis;; Intima-media thickness;; Regression;; Quantitative Coronary Angiography;; Intravascular Ultrasound;; Virtual Histology;; Plaque;; Atorvastatin;
MeSH Terms: conditions — Atherosclerosis; Coronary Disease; Carotid Artery Diseases; Coronary Artery Disease; Plaque, Amyloid | interventions — Blood Component Removal; Apolipoproteins A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Specific Lp(a) apheresis & Atorvastatin (Experimental): Specific Lp(a) apheresis was performed with "Lp(a) Lipopak" immunosorbent columns ("POCARD" Ltd., Moscow, Russia) with sheep polyclonal monospecific antibodies against human Lp(a)/apo(a) weekly during 18 months. On the background - standard medical therapy in accordance with the recommendations for secondary prevention of CHD.
  Interventions: Procedure: Specific Lp(a) apheresis
- Atorvastatin (No Intervention): Standard medical therapy in accordance with the recommendations for secondary prevention of CHD

INTERVENTIONS:
Procedure: Specific Lp(a) apheresis — Specific Lp(a) apheresis procedures were carried out weekly with "Lp(a) Lipopak" columns (POCARD Ltd., Moscow, Russia) according to the standard protocol
  Other Names: "Lp(a) Lipopak" immunoadsorption columns
  Arms: Specific Lp(a) apheresis & Atorvastatin

SUMMARY:
To evaluate whether specific lipoprotein(a) apheresis on the top of optimal medical therapy could affect atherosclerotic disease burden in coronary and carotid arteries of coronary heart disease patients with elevated Lp(a) levels.

DETAILED DESCRIPTION:
Following the hypothesis that if Lp(a) excess has a pathogenic role in atherogenesis, then specific elimination of circulating Lp(a) should affect plaque growth and stability, we evaluated the efficacy of Lp(a) apheresis on changes in coronary plaque volume and composition and carotid intima-media thickness in patients with CHD on the background of optimal medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary heart disease (CHD) requiring a clinically indicated coronary angiography.
* Lp(a) ≥50 mg/dL
* LDL-C <2.6 mmol/L (100 mg/dL)
* Signed written informed consent form to participate in the study

Exclusion Criteria:

* history of acute coronary syndrome or surgical intervention within prior 3 months to inclusion
* chronic infectious and inflammatory diseases
* familial hypercholesterolemia
* TG ≥4.5 mmol/L (400 mg/dL)
* Active liver disease (ALT or AST >3 upper limit of normal (ULN), or total bilirubin >1.5 ULN);
* CK ≥3 ULN;
* Thyroid dysfunction;
* Renal dysfunction (creatinine clearance (Cockcroft-Gault Equation) ≤30 ml/min);
* Uncontrolled diabetes (HbA1c ≥7.0%);
* Coagulopathies;
* Lipid-lowering drugs, except statins for the last month
* Known statin or immunoadsorption intolerance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in Percent Diameter Stenosis | From Baseline to End of Study (Week 72)
  The absolute change from baseline to 18 months in mean percent diameter stenosis, determined by quantitative coronary angiography (QCA) as the narrowest lesion in each segment and calculated as: ((reference diameter-minimal lumen diameter (MLD))/reference diameter)x100.

SECONDARY OUTCOMES:
Change in mean carotid intima-media thickness (IMT) | From Baseline to Week 36 (9 months) and to Week 72 (18 months)
  Change from baseline in mean carotid IMT, as measured by duplex ultrasonography of common carotid arteries after 9 and 18 months.
Numbers of Coronary segments Showing Regression | From baseline to End of study (Week 72)
  Clinically relevant regression or progression was defined as a change from baseline to follow up of ≥10% for percent diameter stenosis
Number of Carotid Segments showing Regression | From Baseline to End of study (Week 72)
  Carotid IMT progression criterion for the 18 months of treatment was considered as growth rate of 0.02 mm (0.015 mm/yr). No changes or reduction in carotid IMT ≥ 0,02 mm served as criterion of stabilization and regression of carotid atherosclerosis, respectively.
Change in total atheroma volume (TAV) from baseline to 18 months post-therapy | From Baseline to Week 72
  TAV at baseline - TAV at Week 72 assessed by intravascular ultrasound (IVUS) imaging of a targeted coronary artery
Change in absolute volumes of plaque components | From Baseline to Week 72
  Mean change in absolute volumes of plaque components: fibrotic, fibrofatty, necrotic core or dense calcium, assessed by radiofrequency intravascular ultrasonographic (IVUS) imaging at baseline and 18 months post-therapy
Change in relative amount of plaque components | From baseline to Week 72
  Mean change in relative amounts of plaque components: fibrotic, fibrofatty, necrotic core or dense calcium, assessed by radiofrequency intravascular ultrasonographic (IVUS) imaging at baseline and 18 months post-therapy
Numbers of Coronary Plaques Showing Regression | From baseline to End of study (Week 72)
  Regression was defined as decrease in TAV for all anatomically comparable cross sectional areas of targeted coronary artery from baseline of ≥ 0,1 mm cubed
Acute change in Lp(a) level | Once a week over 72 week period of active treatment
  Difference in Lp(a) concentration before and after specific Lp(a) apheresis procedure calculated as the mean of all measurements
Change in quality of life (QOL) | from baseline to week 72
  To evaluate the impact of the specific Lp(a) removal therapy on the quality of life using Seattle Angina Questionnaire (SAQ) and Exercise stress test as compared with standard guideline-driven medical therapy of CHD patients

OTHER OUTCOMES:
Total Cholesterol (TC) Serum Level | From Baseline to Week 4, 36, 72
  Mean changes in TC level over the 18-month study period
Lipoprotein(a) (Lp(a)) serum levels | From Baseline to Week 4, 36, 72
  Mean changes in Lp(a) level over the 18-month study period
Low-density lipoprotein cholesterol (LDL-C) serum Level | From Baseline to Week 4, 36, 72
  Mean changes in LDL-C level over the 18-month study period
Change in corrected LDL-C (LDL-C corr) Serum level | From Baseline to Week 4, 36, 72
  Since all included patients had high Lp(a) levels, to avoid overestimation of LDL-C fraction estimated LDL-C levels were corrected for cholesterol derived from Lp(a).
  Corrected LDL-C (LDL-C corr) was calculated using Dahlen's modification of the Friedewald formula: LDL-C corr = TC - (HDL-C) - (TG / 2.2) - (0.3 x Lp(a) / 38.7).
  For values in mmol/L, Lp(a) in mg/dL
Change in triglycerides (TG) serum Level | From Baseline to Week 4, 36, 72
  Mean changes in TG level over the 18-month study period
Change in high-density lipoprotein cholesterol (HDL-C) serum level | From Baseline to Week 4, 36, 72
  Mean changes in HDL-C level over the 18-month study period
Change in hemoglobin level | From Baseline to Week 4, 36, 72
Change in creatinine level | From Baseline to Week 4, 36, 72
Change in creatine kinase (CK) level | From Baseline to Week 4, 36, 72
Change in alanine transaminase (ALT) level | From Baseline to Week 4, 36, 72
Change in aspartate transaminase (AST) level | From Baseline to Week 4, 36, 72

CONTACTS AND LOCATIONS:
Overall Officials: Sergei Pokrovsky, PhD, DSc, Principal Investigator — Russian Cardiology Research and Production Center
Locations (1):
- Russian Cardiology Research and Production Center, Moscow, Russia

REFERENCES:
- [Result] Safarova MS, Ezhov MV, Afanasieva OI, Matchin YG, Atanesyan RV, Adamova IY, Utkina EA, Konovalov GA, Pokrovsky SN. Effect of specific lipoprotein(a) apheresis on coronary atherosclerosis regression assessed by quantitative coronary angiography. Atheroscler Suppl. 2013 Jan;14(1):93-9. doi: 10.1016/j.atherosclerosissup.2012.10.015. PMID 23357149
- [Derived] Pokrovsky SN, Afanasieva OI, Safarova MS, Balakhonova TV, Matchin YG, Adamova IYU, Konovalov GA, Ezhov MV. Specific Lp(a) apheresis: A tool to prove lipoprotein(a) atherogenicity. Atheroscler Suppl. 2017 Nov;30:166-173. doi: 10.1016/j.atherosclerosissup.2017.05.004. Epub 2017 May 31. PMID 29096833
- [Derived] Pokrovsky SN, Afanasieva OI, Ezhov MV. Lipoprotein(a) apheresis. Curr Opin Lipidol. 2016 Aug;27(4):351-8. doi: 10.1097/MOL.0000000000000319. PMID 27213629
- [Derived] Ezhov MV, Safarova MS, Afanasieva OI, Pogorelova OA, Tripoten MI, Adamova IY, Konovalov GA, Balakhonova TV, Pokrovsky SN. Specific Lipoprotein(a) apheresis attenuates progression of carotid intima-media thickness in coronary heart disease patients with high lipoprotein(a) levels. Atheroscler Suppl. 2015 May;18:163-9. doi: 10.1016/j.atherosclerosissup.2015.02.025. PMID 25936321